CLINICAL TRIAL: NCT06411002
Title: A Phase 2a Study to Evaluate the Effects of DaxibotulinumtoxinA for Injection on the Treatment of Dynamic Forehead Lines and Glabellar Lines
Brief Title: Phase 2a Study of DaxibotulinumtoxinA-lanm for Injection in Dynamic Forehead Lines and Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2320201
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Glabellar Frown Lines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active Treatment (DAXXIFY) (Experimental): All subjects will receive DAXXIFY for injection as IM injections.
  Interventions: Drug: DAXXIFY

INTERVENTIONS:
Drug: DAXXIFY — Intramuscular injection of daxibotulintoxinA-lanm
  Other Names: DAXI

SUMMARY:
This is a Phase 2a open-label, single-arm study to evaluate the effects of DaxibotulinumtoxinA-lanm (DAXI) for Injection on the treatment of dynamic forehead lines (FHL) and glabellar lines (GL).

Approximately 40 subjects (18 years of age and above) with moderate to severe GL and FHL (all assessed at maximum contraction) will be screened for eligibility with the goal of enrolling and treating 30 subjects to receive DAXI for injection after providing informed consent.

The primary objective of this study is to determine the efficacy and safety of the combined treatment of two upper facial regions with DAXI for injection.

ELIGIBILITY:
Inclusion Criteria:

1. Be outpatient, male or female subjects, in good general health, 18 years of age or older
2. Have a score of moderate (2) or severe (3) GL during maximum contraction as assessed by the IGA-FWS
3. Have a score of moderate (2) or severe (3) FHL during maximum contraction as assessed by the IGA-FHWS

Exclusion Criteria:

1. Previous treatment with botulinum toxin type A in the face, or treatment with >200 U of any botulinum toxin anywhere else in the body, in the past 6 months prior to screening
2. Pregnant, nursing, or planning a pregnancy during the study; or is a WOCBP but is not willing to use an effective method of contraception
3. Allergy or sensitivity to any botulinum toxin preparations or to any component of the investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
IGA-FWS | Week 4
  • The proportion of subjects achieving a score of 0 (none) or 1 (mild) in GL severity at maximum contraction (maximum frown) at Week 4 as assessed by the IGA-FWS
IGA-FHWS | Week 4
  • The proportion of subjects achieving a score of 0 (none) or 1 (mild) in FHL severity at maximum contraction (maximum eyebrow elevation) at Week 4 as assessed by the IGA-FHWS

CONTACTS AND LOCATIONS:
Locations (1):
- Revance, Nashville, Tennessee, United States